CLINICAL TRIAL: NCT02519179
Title: Influence of Bottle-Type of Infant Feeding Behavior
Acronym: OBS-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California Polytechnic State University-San Luis Obispo (Other)
Responsible Party: Principal Investigator, Alison Ventura, Assistant Professor, California Polytechnic State University-San Luis Obispo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 00000
Record Dates: First submitted 2015-08-05; First posted 2015-08-10 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-01

CONDITIONS: Bottle Feeding
MeSH Terms: conditions — Bottle Feeding

STUDY DESIGN:
Intervention Model Description: This is a within-subject study; mothers are observed during both feeding conditions.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Conventional vs. Opaque, Weighted Bottle (Experimental): This is a within-subject experiment; mothers will be asked to feed their infants from a clear, conventional bottle during one visit and an opaque, weighted bottle during the other visit. Order of conditions will be counterbalanced.
  Interventions: Behavioral: Opaque, weighted bottle; Behavioral: Clear, conventional bottle

INTERVENTIONS:
Behavioral: Opaque, weighted bottle — This is the experimental condition; mothers will be asked to feed their infants from an opaque, weighted bottle.
Behavioral: Clear, conventional bottle — This is the control condition; mothers will be asked to feed their infants from a clear, conventional bottle.

SUMMARY:
The objective this research is to conduct a within-subject, experimental study that will describe mothers' feeding practices during typical bottle-feeding conditions and will examine whether removal of visual cues related to the amount of milk/formula in the bottle will alter these feeding practices. The investigators hypothesize that mothers will show higher levels of infant-directed feeding practices and lower levels of mother-directed feeding practices when using opaque, weighted bottles compared to when using standard, clear bottles. The investigators also hypothesize that infants will consume less breast milk or formula when fed from opaque, weighted bottles compared to when fed from standard, clear bottles.

ELIGIBILITY:
Inclusion Criteria:

* Mothers must be 18 years or older
* Infants must be between 0-6 months of age
* Infants must be prior to the introduction of solid foods

Exclusion Criteria:

* Preterm birth
* Medical conditions that interfere with feeding

Max Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Infant intake | 3-hour period
  Infant intake within a feeding (mL) assessed by weighing the bottle before and after a feeding.
Maternal responsiveness | 3-hour period
  Maternal responsiveness to infant cues during a feeding assessed by Nursing Child Assessment Satellite Training Parent-Child Interaction Feeding Scale.

SECONDARY OUTCOMES:
Maternal acceptance/perception of intervention | 3-hour period
  Maternal perception/acceptance of the bottles during a feeding assessed through a mixed methods interview.

CONTACTS AND LOCATIONS:
Overall Officials: Alison K Ventura, PhD, Principal Investigator — Assistant Professor
Locations (1):
- California Polytechnic State University, San Luis Obispo, California, United States

REFERENCES:
- [Background] Ventura AK, Pollack Golen R. A pilot study comparing opaque, weighted bottles with conventional, clear bottles for infant feeding. Appetite. 2015 Feb;85:178-84. doi: 10.1016/j.appet.2014.11.028. Epub 2014 Nov 28. PMID 25445988